CLINICAL TRIAL: NCT01439321
Title: Outcomes Comparison of Chronic Immune Thrombocytopenic Purpura (ITP) Patients Switched to Eltrombopag and Romiplostim
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113922
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: treatment satisfaction; romiplostim; eltrombopag; chronic immune thrombocytopenic pupura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; romiplostim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with Chronic Immune Thrombocytopenic Purpura: Patients with chronic ITP who switch from their previous treatment of corticosteroids, rituximab, or eltrombopag or romiplostim to eltrombopag or romiplostim and have been on the new treatment for at least four weeks
  Interventions: Biological: Eltrombopag; Biological: Romiplostim

INTERVENTIONS:
Biological: Eltrombopag — Switched to Eltrombopag
  Other Names: Promacta® is a registered trademark of GlaxoSmithKline
Biological: Romiplostim — Switched to Romiplostim
  Other Names: Nplate® is a registered trademark of Amgen

SUMMARY:
Chronic immune thrombocytopenic purpura (ITP) is characterized by low platelet counts and the risk of severe bleeding complications. The two recently introduced TPO-RA drugs, namely, eltrombopag and romiplostim, have shown efficacious sustained response with continuous administration. Both drugs are indicated for the treatment of thrombocytopia in patients with chronic ITP who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy. While these trials address important clinical questions they were not intended to evaluate what happens in the real-world settings with actual patient living daily lives. The purpose of this health outcomes study is to understand how the two TPO receptor agonists (TPO-RA) currently available in the US are being used in clinical practice and how their use impacts chronic ITP patients' daily lives. The study hypothesis is that patients who switched to eltrombopag report a better health-related quality of life than those who switched to romiplostim. This study utilized a hybrid design of retrospective chart review study and cross-sectional patient survey. A customized Patient Case Report Form (CRF) will be used to retrospectively collect clinical data from patient medical charts where the primary cohorts consist of patients who have switched from other ITP medication to eltrombopag or romiplostim. A cross-sectional survey will be employed to collect patient reported outcomes (PRO) data, including health-related quality of life and treatment satisfaction, using a compository questionnaire. Analyses of cross-sectional survey data and retrospective medical chart review data in patients who switch to either eltrombopag or romiplostim from their prior primary therapy will be conducted.

ELIGIBILITY:
Inclusion criteria

* Adults 18 years and older diagnosed with chronic ITP
* Switched to eltrombopag or romiplostim a minimum of 4 weeks prior to index date
* Received corticosteroids, rituximab, or one TPO-receptor agonist as prior primary therapy before switching to eltrombopag or romiplostim
* Medical history must be available from chronic ITP diagnosis through to most recent office visit
* Patients who complete the self-administered questionnaire were the same patients whose medical charts were reviewed

Exclusion criteria

* Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include adult patients with a diagnosis of immune (idiopathic) thrombocytopenic purpura (ITP) who switched to eltrombopag or romiplostim.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
treatment satisfaction scores by domain | During a 5 month period, the questionnaire will be administered to each participant at one time point. The recall period for the TQSM in this study is 3 weeks
  Treatment satisfaction will be captured with the Treatment Satisfaction Questionnaire for Medication (TSQM). The questionnaire is composed of 14 items. Mean scores will be reported for each treatment group by domain. The domains of the TSQM are effectiveness, side effects, convenience, and global satisfaction

SECONDARY OUTCOMES:
Short-form 36 (SF-36) score | During a 5 month period, the questionnaire will be administered to each participant at one time point. The recall period for the SF-36 in this study is 1 week
  The SF-36 is a general overall health instrument consisting of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Scales include general health, limitations of activities, physical functioning, emotional health, social activities, pain, and energy/ emotional functioning. Scores for social functioning and physicial functioning will also be reported

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline